CLINICAL TRIAL: NCT03342534
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Brain Organization and Motor Recovery After Stroke
Brief Title: Effect of tDCS on Brain Organization and Motor Recovery
Acronym: ESTCORM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of funds before obtaining the planned number of patients.
Sponsor: Adrian Guggisberg (Other)
Collaborators: University Hospital, Geneva (Other); Clinique Romande de Readaptation (Network); Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Sponsor-Investigator, Adrian Guggisberg, Médecin adjoint agrégé, assistant professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRSII5-170985A
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Anodal tDCS (Active Comparator): The anode is placed over the primary motor cortex of the stroke affected hemisphere, the cathode over the contralesional supraorbital front of the patient.
  Interventions: Device: DC-stimulator (Neuroconn, Germany)
- High definition (HD) anodal tDCS (Active Comparator): A single HD anode is placed over the primary motor cortex of the stroke affected hemisphere, 4 HD cathodes are placed over the affected hemisphere around the anode.
  Interventions: Device: DC-stimulator (Neuroconn, Germany)
- Bihemispheric tDCS (Active Comparator): The anode is placed over the primary motor cortex of the stroke affected hemisphere, the cathode over the primary motor cortex of the contralesional hemisphere.
  Interventions: Device: DC-stimulator (Neuroconn, Germany)
- Sham tDCS (Sham Comparator): The electrodes are placed as in one of the active arms, but only a ramp up current is applied during 30 seconds and then switched off. This induces similar sensations for the patients, but no change in excitability.
  Interventions: Device: DC-stimulator (Neuroconn, Germany)

INTERVENTIONS:
Device: DC-stimulator (Neuroconn, Germany) — A current of 2 mA will be applied for 20 minutes, 3 times per week during 2 weeks, except for the sham tDCS arm.

SUMMARY:
Neurological deficits and motor disorders are extremely common after stroke. Physical therapies can improve the autonomy of these patients, but despite an intensive stationary neurorehabilitation, severe deficits often persist. Complementary therapies that could improve recovery would therefore be very welcome.

Transcranial direct current stimulation (tDCS) induces, in a non-invasive way, a transient inhibitory or excitatory neuromodulation of certain cerebral regions. An increasing number of studies show that this modulation of brain activity can improve motor functions in patients with brain lesions and increase the effect of physical therapies. However, the "optimum" configuration of tDCS and the induced effects remain to be characterized and investigated.

The investigators therefore propose to carry out a study including a pilot phase in order to determine the most efficient tDCS setup. The optimum setup of of the pilot phase will be compared to a placebo condition in a multicentric main study.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke
* ≤ 4 weeks after stroke onset
* Paresis of upper limb with Fugl-Meyer score between 15 and 55 at study entry
* Capable of participating during treatment sessions of 30-60 minutes
* Informed consent obtained

Exclusion Criteria:

* Incapacity to understand study information or task instructions during trial.
* New additional stroke during rehabilitation
* Reduced vigilance or delirium
* Severe language deficits
* Preexisting affection of an upper limb
* Severe spasticity or dystonia
* Severe co-morbidities (e.g., traumatic, rheumatologic, neurodegenerative disease)
* Pregnancy
* Pacemaker
* Skull breach
* History of seizures or epilepsy
* Metallic object in the brain
* Other contraindication to non-invasive brain stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in upper extremity Fugl-Meyer score, after intervention | Difference between the week before the intervention and the week after intervention
  Scale range 0-66 points, higher values indicate better outcome. Assessed by qualified physical or occupational therapists

SECONDARY OUTCOMES:
Change in EEG functional connectivity, after intervention | Difference between the week before the intervention and the week after intervention
  EEG functional connectivity between ipsilesional motor cortex and the rest of the brain, as computed from high-density EEG recordings. Continuous measure. Higher values indicate better outcome.
Change in amplitude of motor evoked potentials, after intervention | Difference between the week before the intervention and the week after intervention
  Motor evoked potentials are obtained with single-pulse transcranial magnetic stimulation. Continuous measure expressed in microvolts, more microvolts indicate better outcome.

OTHER OUTCOMES:
Change in upper extremity Fugl-Meyer score, follow up 1 | Difference between the week before intervention and 4 weeks after intervention
  Scale range 0-66 points, higher values indicate better outcome. Assessed by qualified physical or occupational therapists
Change in upper extremity Fugl-Meyer score, follow up 2 | Difference between the week before intervention and 12 weeks after stroke onset
  Scale range 0-66 points, higher values indicate better outcome. Assessed by qualified physical or occupational therapists
Change in Jamar dynamometer, after intervention | Difference between the week before the intervention and the week after intervention
  Continous measure expressed in kilograms. Higher values indicate better outcome. Assessed by qualified physical or occupational therapists
Change in Jamar dynamometer, follow up 1 | Difference between the week before intervention and 4 weeks after intervention
  Continous measure expressed in kilograms. Higher values indicate better outcome. Assessed by qualified physical or occupational therapists
Change in Jamar dynamometer, follow up 2 | Difference between the week before intervention and 12 weeks after stroke onset
  Continous measure expressed in kilograms. Higher values indicate better outcome. Assessed by qualified physical or occupational therapists
Change in Nine-Hole-Peg test, after intervention | Difference between the week before the intervention and the week after intervention
  Expressed in pegs/second. Higher values indicate better outcome. Assessed by qualified physical or occupational therapists.
Change in Nine-Hole-Peg test, follow up 1 | Difference between the week before intervention and 4 weeks after intervention
  Expressed in pegs/second. Higher values indicate better outcome. Assessed by qualified physical or occupational therapists.
Change in Nine-Hole-Peg test, follow up 2 | Difference between the week before intervention and 12 weeks after stroke onset
  Expressed in pegs/second. Higher values indicate better outcome. Assessed by qualified physical or occupational therapists.
Change in action research arm test (ARAT) score, after intervention | Difference between the week before the intervention and the week after intervention
  Scale range 0-57 points, higher values indicate better outcome. Assessed by qualified physical or occupational therapists
Change in action research arm test (ARAT) score, follow up 1 | Difference between the week before intervention and 4 weeks after intervention
  Scale range 0-57 points, higher values indicate better outcome. Assessed by qualified physical or occupational therapists
Change in action research arm test (ARAT) score, follow up 2 | Difference between the week before intervention and 12 weeks after stroke onset
  Scale range 0-57 points, higher values indicate better outcome. Assessed by qualified physical or occupational therapists
Change in Functional Independence Measure (FIM) score, after intervention | Difference between the week before the intervention and the week after intervention
  Range 18-126, higher values indicate better outcome. Assessed by rehabilitation nurses.
Change in Functional Independence Measure (FIM) score, follow up 1 | Difference between the week before intervention and 4 weeks after intervention
  Range 18-126, higher values indicate better outcome. Assessed by rehabilitation nurses.
Change in Functional Independence Measure (FIM) score, follow up 2 | Difference between the week before intervention and 12 weeks after stroke onset
  Range 18-126, higher values indicate better outcome. Assessed by rehabilitation nurses.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian G Guggisberg, MD, Principal Investigator — University of Geneva; José Millán, PhD, Study Director — University of Texas at Austin
Locations (2):
- Switzerland (2):
  - Division of Neurorehabilitation, University Hospital of Geneva, Geneva, Canton of Geneva
  - Universitäre Neurorehabilitation, Inselspital, Bern